CLINICAL TRIAL: NCT02649127
Title: The Role of Exercise in the Treatment of PTSD
Brief Title: The Role of Exercise in the Treatment of PTSD Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: C.R.Darnall Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC20100372H
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2016-09

CONDITIONS: Posttraumatic Stress Disorder
Keywords: exercise; biomarker
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity | interventions — Implosive Therapy; Exercise; Self Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Imaginal Therapy Only (Experimental): The imaginal exercise of exposure therapy will be manualized (Rothbaum, Foa & Hembree, 2007) and adapted with the permission of Dr. Foa for combat-related stress disorders (Peterson, Cigrang & Riggs, 2008). While traditional exposure therapy includes both imaginal exposure and in vivo exposure, this study will use only the imaginal exposure components. Participants will meet with a therapist the first week of treatment and every-other week for a total of five appointments over eight weeks. During the second session, the therapist will help the participant make an approximately 20-minute voice tape recording of their traumatic experience which they will listen to 5-days/week. A new recording will be made with the therapist during sessions 3 and 4 also, for a total of three tapes.
  Interventions: Behavioral: imaginal therapy
- Exercise Only (Experimental): The aerobic exercise regimen will be standardized according to the American College of Sports Medicine recommendations: frequency of a minimum of 5 sessions per week, at a vigorous intensity [>60% of oxygen uptake reserve (VO2R)], time of 20-25 minutes per exercise session. To determine the exercise heart rate intensity, the Karvonen formula for heart rate reserve will be used. The mode of exercise will be purposeful walking or jogging. The goal of the exercise is not training, but rather to keep the participant's heart rate >60% of their individually-determined heart rate reserve.
  Interventions: Behavioral: exercise
- Imaginal Therapy & Exercise Combined (Experimental): Participants will meet with a therapist the first week of treatment and every-other week for a total of five appointments over eight weeks. During the second session, the therapist will help the participant make an approximately 20-minute voice tape recording of their traumatic experience which they will listen to 5-days/week. A new recording will be made with the therapist during sessions 3 and 4 also, for a total of three tapes. Participants will exercise listening to their tape at least 5-times/week outside of scheduled unit Physical Training. Participants will wear the heart rate monitor to record their exercise activity.
  Interventions: Behavioral: imaginal therapy; Behavioral: exercise
- Nurse-led Self-Care (Active Comparator): The Self-Care Group will use written materials that outline the benefits of thinking about problems the individual is facing as well as the benefits of exercise, however doing the two activities together will not be advocated as part of the material. A fact sheet prepared by the National Center for PTSD, Returning from the War Zone: A Guide for Military Personnel as well as a list of coping strategies and self-care behaviors adapted from the National Center for PTSD guide, Self-Care and Self-Help Following Disasters, will be used to guide the discussion. The research nurse will meet with the participant five times over 8-weeks at weeks 1, 2, 4, 6, and 8 to encourage use of the self-care fact sheet and assess the participant for safety.
  Interventions: Behavioral: self-care

INTERVENTIONS:
Behavioral: imaginal therapy — imaginal exercise of Prolonged Exposure therapy
  Arms: Imaginal Therapy & Exercise Combined; Imaginal Therapy Only
Behavioral: exercise — aerobic training at a frequency of a minimum of 3 sessions per week, at vigorous intensity [i. e., >60% of oxygen uptake reserve (VO2R)], and a time of 20-25 minutes each bout of training
  Arms: Exercise Only; Imaginal Therapy & Exercise Combined
Behavioral: self-care — meeting with a nurse to review and discuss publically available written materials that outline approaches for dealing with posttraumatic stress symptoms
  Arms: Nurse-led Self-Care

SUMMARY:
This is an 8-week experimental, repeated-measures clinical trial randomizing 120 Service Members with symptoms of PTSD into one of four groups: 1) imaginal exercises of exposure therapy only, 2) aerobic exercise only, 3) imaginal exercises augmented with aerobic exercise, or 4) self-care.

DETAILED DESCRIPTION:
One of the signature injuries of combat operations following 9/11 is posttraumatic stress disorder (PTSD). The most effective treatment for PTSD is exposure therapy where, under the supervision of a trained therapist, individuals are exposed to prolonged and repeated imagined images of the trauma until the images no longer cause severe anxiety. Various forms of exercise have been used to treat a broad range of depression and anxiety disorders and exercise has been used with some success to treat individuals with PTSD. Considering the population of otherwise healthy and physically active Service Members suffering from symptoms of PTSD, it seems possible that exercise might serve as an outlet for the emotional reactions experienced during therapy, decreasing emotional distress, and increasing the individual's tolerance to imaginal exposure serving as a powerful adjunct to exposure therapy. The purpose of this study to explore the role of exercise in the treatment of symptoms of posttraumatic stress disorder (PTSD), specifically determining if the efficacy of imaginal exercises, part of exposure therapy for PTSD, can be improved by augmenting the therapy with aerobic exercise. Towards this end, this 8-week experimental, repeated-measures clinical trial will randomize 120 Service Members with symptoms of PTSD into one of four groups: 1) imaginal exercises of exposure therapy only, 2) aerobic exercise only, 3) imaginal exercises augmented with aerobic exercise, or 4) self-care.

ELIGIBILITY:
Inclusion Criteria:

* be an Active Duty, Reserve, or National Guard Army, Air Force, Navy, or Marine Veteran of Operation Iraqi Freedom (OIF) / Operation Enduring Freedom (OEF) eligible for military medical care
* be at least 18 years old
* be able to read and speak English
* answer "no" to the seven questions of the Physical Activity Readiness Questionnaire (PAR-Q), or have primary care provider approval to undertake an exercise program.
* score ≥25 on the PTSD CheckList - Stressor-Specific(PCL-S); participants scoring >50 on the PCL-S will be contacted weekly to ensure that their symptoms are under control and they do not require a higher level of care.
* report on the PTSD Symptom Scale - Interview (PSS-I) an exposure to a traumatic event (Criterion A), at least one re-experiencing symptom (Criterion B), and at least one avoidance symptom (Criterion C)
* participants taking psychotropic medications agree to work with their prescriber to remain on stable doses of any prescribed psychotropic medications for the duration of the intervention and through the 1-month follow-up assessment as much as possible and as medically indicated
* anticipate being in the area for at least three months to complete intervention and 13-week follow-up assessment

Exclusion Criteria:

* score <25 on the PTSD CheckList - Stressor Specific (PCL-S) (Those scoring <25 do not have enough symptom severity to adequately test the study hypotheses
* have undergone exposure therapy for PTSD within the last year
* be taking benzodiazepines every day on a prescribed schedule (Individuals prescribed and taking a benzodiazepine only as needed will not be excluded.)
* suicidal ideation with moderate to severe intent warranting intervention
* active psychosis or mania
* be on a medical profile that prohibits exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms as assessed using the PTSD Symptom Scale - Interview (PSS-I) and PTSD CheckList (PCL) | change in score between baseline, 1-week post-treatment, 1-month post-treatment, 6-months post-treatment
  degree of PTSD symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Young-McCaughan, RN, PhD, Principal Investigator — University of Texas Health Science Center San Antonio
Locations (1):
- Carl R. Darnall Army Medical Center, Fort Hood, Texas, United States

REFERENCES:
- See also: STRONG STAR Consortium web link describing study — http://tango.uthscsa.edu/strongstar/subs/afinfo.asp?prj=17